CLINICAL TRIAL: NCT00491075
Title: Phase II Trial of Pemetrexed Plus Gemcitabine in Patients With Advanced Non-Clear Cell Renal Cell Cancer
Brief Title: Pemetrexed Plus Gemcitabine in Renal Cell Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed early for poor accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0516
Record Dates: First submitted 2007-06-21; First posted 2007-06-25 (Estimated); Results first posted 2012-05-03 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal Cell Carcinoma; Non-Clear Cell; Pemetrexed; Gemcitabine; LY231514; Alimta; MTA; Multitargeted Antifolate; NSC-698037; Gemcitabine Hydrochloride; Gemzar; RCC
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Pemetrexed; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pemetrexed + Gemcitabine (Experimental): Pemetrexed 500 mg/m^2 intravenous (IV) and Gemcitabine 1500 mg/m^2 IV on Day 1.
  Interventions: Drug: Pemetrexed; Drug: Gemcitabine

INTERVENTIONS:
Drug: Pemetrexed — 500 mg/m^2 IV Over 10 Minutes on Day 1.
  Other Names: LY231514; Alimta; MTA; Multitargeted Antifolate; NSC-698037
Drug: Gemcitabine — 1500 mg/m^2 IV Over 30 Minutes on Day 1, Immediately After Infusion of Pemetrexed.
  Other Names: Gemcitabine Hydrochloride; Gemzar

SUMMARY:
Primary Objective:

* To determine the clinical activity of Pemetrexed + Gemcitabine in non-clear cell renal cell cancer (RCC). Clinical activity will take into account response rate and progression free survival (PFS).

Secondary Objectives:

* To determine the toxicity of Pemetrexed + Gemcitabine in non-clear cell RCC.
* To estimate the survival rate of patients with non-clear cell RCC treated with this combination.

DETAILED DESCRIPTION:
Pemetrexed is a chemotherapy drug that is used to treat cancer. It is given intravenously (by IV--through a vein in your arm). It interferes with cell reproduction.

Gemcitabine is a cancer-fighting (chemotherapy) drug that is given by IV. It interferes with the growth of cells and is used to treat cancer.

Dexamethasone has many different medical uses. It is used to treat cancer, nausea, vomiting, inflammation, allergic reactions, and many other conditions. In this study, it is being given to prevent rashes.

Folic acid and Vitamin B12 are vitamins given to prevent serious side effects which can occur with chemotherapy. These side effects include diarrhea and a decrease in you red blood cells, white blood cells, and your blood platelets.

You will be required to take folic acid and vitamin B12. You will take folic acid, by mouth, daily beginning about 1 week before the first dose of Pemetrexed. You will continue to take it daily until 3 weeks after the last dose of chemotherapy. Vitamin B12 will be given as an injection into your muscle about 1 to 2 weeks before your first dose of Pemetrexed. You will have injections of vitamin B12 about every 9 weeks until 3 weeks after your last dose of chemotherapy.

During treatment, you will be given Pemetrexed by IV for 10 minutes, followed by Gemcitabine by IV for 30 minutes on Day 1 of each 2-week study "cycle."

You will take Dexamethasone tablets by mouth, 2 times a day on the day before, the day of, and the day after each dose of Pemetrexed. Dexamethasone is taken to prevent rashes. If you could not or did not take Dexamethasone the day before and/or the day of Pemetrexed, you may be given Dexamethasone by IV over 20 minutes, 30 minutes before the infusion of Pemetrexed.

You will have blood samples (about 4 teaspoons) drawn every week to test your bone marrow. You will have blood samples (about 1 teaspoon) drawn every 2 weeks to make sure that your kidneys and liver are working well. You will have a physical exam every 2 weeks before you receive chemotherapy. You will also be asked about any medications you have been taking since your last visit.

Once every 8 weeks or after 4 cycles of treatment, you will have the tumor(s) measured using standard of care imaging which may include a CT scan, MRI, or a bone scan.

You will be treated for as long as you are benefiting from the therapy. You will continue to receive treatment unless your tumor grows, intolerable side effects occur, or you develop another illness that prevents you from continuing with the therapy. You may also be taken off study if you fail to comply with the study requirements. If you are taken off study for any reason, you and your doctor will discuss other treatment options at that time.

If you are taken off study, you will be asked to have the same scans as before, a physical exam, and routine blood (about 4 teaspoons). You will be contacted every 3 months after being off study, to get an update on your health status.

This is an investigational study. Pemetrexed and Gemcitabine are FDA approved and commercially available. About 40 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed advanced non-clear cell RCC. Patients with locally recurrent disease are eligible. Patients with locally advanced unresectable RCC should have measurable metastatic disease to be eligible for the protocol. Patients with bilateral renal cancer are eligible as long as both cancers are of non-clear cell type and patients have metastatic disease.
* Patients must have measurable disease.
* Patients with previously treated or untreated, non-threatening brain metastasis are eligible. For previously treated patients, prior whole brain radiation therapy or stereotactic radiosurgery must be > 3 months from initiation of current therapy and there can be no plans for concurrent radiation while on this study. Patients who had surgical resection for brain metastasis are eligible to enroll after they recover from surgery.
* Life expectancy > 8 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Patients must have adequate organ and marrow function as defined below: (1) Hemoglobin >/= 9g/dl; (2) absolute neutrophil count >/= 1,500/microL; (3) platelets >/=100,000/microL; (4) total bilirubin </= 1.5 mg/dl; (5) aspartate aminotransferase (AST or SGOT) and/or alanine aminotransferase (ALT or SGPT) (SGPT) </= 2.5 * institutional upper limits of normal (uln), or </= 5 * uln if liver metastasis exists; (6) creatinine clearance (calculated by the Cockcroft-Gault formula) >/= 45 mL/min
* Patients must have recovered from any effects of surgery and/or radiation therapy and be free of significant detectable infection.
* Female patients of childbearing potential must have a normal plasma beta human chorionic gonadotropin (bHCG) within 24 hours prior to enrolling in the study. Patients with an elevated bHCG will undergo appropriate evaluation to rule out pregnancy (ie referral to OB-Gyn service, ultrasound) and if pregnancy is ruled out and elevated bHCG is determined to be of tumor origin, patients will be permitted to proceed on study.
* Patients of child fathering or childbearing potential must agree to practice a form of medically acceptable birth control while on study
* Patients must give written consent prior to initiation of therapy, in keeping with the policies of the institution. Patients with a history of major psychiatric illness must be judged able to fully understand the investigational nature of the study and the risks associated with the therapy. The only approved consent is attached to this protocol.

Exclusion Criteria:

* Pregnant or lactating women.
* No prior malignancy is allowed, except for non-melanoma skin cancer, in situ carcinoma of any site, or other cancers for which the patient has been adequately treated and disease free for 2 years.
* Patients must not have received more than 2 prior systemic therapies for RCC, but patients should not have received any prior chemotherapy for RCC. Chemotherapy given for other types of cancer more than 2 years prior to enrollment on this protocol is permitted.
* Patients must not be scheduled to receive any experimental drug for MRCC while on study. Patients are permitted to be on concomitant bisphosphonates or megestrol acetate. Patients are permitted to receive hematopoietic growth factors according to American Society of Clinical Oncology (ASCO) guidelines.
* Patients must not have had prior radiotherapy to areas of measurable disease, unless they have clearly progressive disease in this site, or there is measurable disease outside the area of prior radiation. Radiotherapy, if needed for palliation, must have been completed prior to enrollment on this study.
* Patients must not have any significant medical disease (other than the malignancy) that, in the opinion of the investigator, would significantly increase the risk for participation in this trial. Examples of exclusion: unstable angina pectoris, New York Heart Association (NYHA) Grade II or greater congestive heart failure, unstable symptomatic cardiac arrhythmias requiring medication (subjects with controlled chronic atrial fibrillation are eligible), myocardial infarction within the last 6 months, uncontrolled hypertension (blood pressure >160/110 on therapy) or uncontrolled diabetes mellitus.
* Patients must not have history of other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications.
* Patients unwilling to participate or unable to comply with the protocol for the duration of the study.
* Inability or unwillingness to take corticosteroid, folic acid or vitamin B12 supplementation.
* Inability to interrupt aspirin or other non-steroidal anti-inflammatory agents for a 5 day period (for short acting NSAIDs) or 8-day period (for long-lasting NSAIDs, such as piroxicam)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2005-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nizar M. Tannir, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD . Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Background] Richey SL, Tamboli P, Ng CS, Lin E, Lim ZD, Araujo JC, Jonasch E, Sharma P, Pagliaro LC, Tannir NM. Phase II trial of pemetrexed plus gemcitabine in patients with locally advanced and metastatic nonclear cell renal cell carcinoma. Am J Clin Oncol. 2013 Oct;36(5):450-4. doi: 10.1097/COC.0b013e3182546a91. PMID 22706175

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: December 13, 2005 through January 02, 2009. Participants were recruited from the UT MD Anderson's Genitourinary (GU) Cancer Center medical clinic.
Period: Overall Study
Arm/Group | Pemetrexed + Gemcitabine
Started | 16
Completed | 14
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed + Gemcitabine
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 54 (12.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Overall Response
Description: Number of participants with complete or partial response. Response Evaluation Criteria in Solid Tumors (RECIST) of Complete Response: disappearance all target lesions; Partial Response: >30% decrease in sum of longest diameter (LD) of target lesions, reference baseline sum LD; Progressive Disease: >20% increase sum of LD of target lesions, reference smallest sum LD recorded since treatment started or appearance of 1 or > new lesions; Stable Disease: Insufficient shrinkage for partial response, or insufficient increase for progressive disease, reference smallest sum LD since treatment started.
Time Frame: Baseline to 8 weeks (after 4 cycles) protocol response at 16 weeks
Population: One participant did not meet the required 16 week data end point and was excluded from the response evaluation and analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed + Gemcitabine
Number analyzed (Participants) | 14
percentage of participants | 6.7 [0.2 to 31.9]

ADVERSE EVENTS:
Time Frame: 3 Years
Description: Of the 16 participants enrolled, one participant started the study but withdrew prior to receiving any treatment and is therefore excluded from adverse event reporting.
Arm/Group | Pemetrexed + Gemcitabine
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed + Gemcitabine (N=15)
thromboembolic event (Vascular disorders) | 1 (1) — Pulmonary embolism
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed + Gemcitabine (N=15)
white blood cell decreased (Investigations) | 8 (8) — leukocytopenia
neutrophil count decreased (Investigations) | 8 (8) — Neutropenia
anemia (Blood and lymphatic system disorders) | 2 (2)
INR increased (Investigations) | 1 (1) — prolonged INR
fatigue (General disorders) | 6 (6)
renal failure (Renal and urinary disorders) | 2 (2)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1)
alanine aminotransferase increased (Investigations) | 1 (1) — ALT or SGPT (serum glutamic pyruvic transaminase) or transaminitis
aspartate aminotransferase (Infections and infestations) | 1 (1) — AST, SGOT (serum glutamic oxaloacetic transaminase) or transaminitis
fever (in the absence of neutropenia) (General disorders) | 1 (1) — non-neutropenic fever

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No